CLINICAL TRIAL: NCT06929325
Title: A Randomized, Double-blind, Multicenter Phase III Clinical Study to Evaluate the Efficacy and Safety of Sirolimus for Injection (Albumin-bound) Combined With Fulvestrant Versus Placebo Combined With Fulvestrant in HR-positive, HER2-negative Locally Advanced or Metastatic Breast Cancer Patients After Prior CDK4/6 Inhibitor Treatment.
Brief Title: Sirolimus for Injection (Albumin-bound) Combined With Fulvestrant for HR+/HER2- Advanced/Metastatic Breast Cancer Patients Previously Treated With CDK4/6 Inhibitors
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HB1901-008
Record Dates: First submitted 2025-04-08; First posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: HR+/HER2- Advanced/Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Sirolimus; Injections; Fulvestrant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sirolimus for Injection (Albumin-bound) Combined with Fulvestrant (Experimental)
  Interventions: Drug: Sirolimus for Injection (Albumin-bound); Drug: Fulvestrant Injection
- Placebo Combined with Fulvestrant (Active Comparator)
  Interventions: Drug: Fulvestrant Injection; Drug: Placebo for Sirolimus for Injection (Albumin-bound)

INTERVENTIONS:
Drug: Sirolimus for Injection (Albumin-bound) — IV infusion, every 2 weeks, 4 weeks per treatment cycle
  Arms: Sirolimus for Injection (Albumin-bound) Combined with Fulvestrant
Drug: Fulvestrant Injection — IM injection, 500 mg, on day 1 and day 15 of Cycle 1, and then on day 1 of each cycle thereafter, 4 weeks per treatment cycle
Drug: Placebo for Sirolimus for Injection (Albumin-bound) — IV infusion, every 2 weeks, 4 weeks per treatment cycle
  Arms: Placebo Combined with Fulvestrant

SUMMARY:
A randomized, double-blind, multicenter phase III clinical study to evaluate the efficacy and safety of sirolimus for injection (albumin-bound) combined with fulvestrant in patients with HR+ and HER2- advanced breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* 1. Aged 18 or above, regardless of gender; female patients must be postmenopausal, or premenopausal/perimenopausal.
* 2. Pathologically confirmed HR+, HER2- breast cancer.
* 3. Locally advanced or metastatic breast cancer, not suitable for curative surgery or radiotherapy, and no current clinical indication for chemotherapy.
* 4. Previously received at least one, up to two lines of systemic therapy (including at least one line of endocrine therapy combined with CDK4/6 inhibitor therapy).
* 5. At least one measurable lesion according to RECIST 1.1 criteria.
* 6. Willing to provide tumor and/or blood samples for biomarker testing; if unable to provide, subject to investigator and sponsor evaluation for eligibility.
* 7. ECOG performance status score of 0-1.
* 8. Investigator-assessed life expectancy ≥6 months.
* 9. Adequate organ and bone marrow function.
* 10. Premenopausal female patients using LHRH agonists to suppress ovarian function must agree to use two acceptable forms of highly effective contraception during the study and for 2 years after stopping study treatment; female patients of childbearing potential must have a negative pregnancy blood test before starting study treatment and must not be breastfeeding.
* 11. Male patients must agree to use barrier contraception (i.e., condoms) during the study and for 2 years after stopping study treatment; for men with future fertility plans, sperm freezing is recommended before starting study treatment.
* 12. Participants must provide informed consent before the trial and voluntarily sign the written ICF.

Exclusion Criteria:

* 1. Previous pathological diagnosis of HER2-positive breast cancer.
* 2. Patients judged by the investigator to be unsuitable for endocrine therapy.
* 3. Patients who have previously received PI3K/AKT/mTOR inhibitors, fulvestrant, or other ER-targeted therapies (including oral SERDs, ER protein degraders PROTAC, etc.).
* 4. Received chemotherapy, radiotherapy, biological therapy, targeted therapy, immunotherapy, or other anti-tumor treatments within 4 weeks before randomization.
* 5. Received other unapproved investigational drugs within 4 weeks before randomization.
* 6. Underwent major surgery within 4 weeks before randomization or has not fully recovered from any previous invasive procedures.
* 7. Received systemic glucocorticoids (prednisone >10 mg/day or equivalent) or other immunosuppressive treatments within 2 weeks before randomization.
* 8. Had an infection within 2 weeks before randomization requiring systemic (oral or IV) anti-infective treatment (uncomplicated urinary tract infections or upper respiratory tract infections excluded).
* 9. Received inactivated or live attenuated vaccines or COVID-19 vaccines within 4 weeks before randomization.
* 10. Used strong inhibitors or inducers of CYP3A4 hepatic metabolic enzymes within 2 weeks before randomization or still need to continue using such drugs.
* 11. Diagnosed with other malignancies within 5 years before randomization.
* 12. Suffering from severe cardiovascular or cerebrovascular diseases.
* 13. Adverse reactions from previous anti-tumor treatments have not recovered to CTCAE 5.0 grade ≤1.
* 14. Active leptomeningeal disease or poorly controlled central nervous system metastases.
* 15. Presence of pleural/abdominal effusion or pericardial effusion with clinical symptoms or requiring symptomatic treatment.
* 16. Known bleeding tendency (constitution) or coagulation disorders.
* 17. History of severe lung diseases such as interstitial lung disease and/or pneumonia, pulmonary hypertension, or radiation pneumonitis requiring glucocorticoid treatment.
* 18. Known hypersensitivity or intolerance to any component of the study drug or its excipients, or LHRH agonists (if applicable).
* 19. History of autoimmune diseases (except tuberous sclerosis), immunodeficiency diseases, including HIV-positive, or other acquired or congenital immunodeficiency diseases, or organ transplant history.
* 20. Active HBV, HCV, syphilis, or tuberculosis infection.
* 21. Other conditions judged by the investigator to be unsuitable for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival（PFS） | Up to ~24 months

SECONDARY OUTCOMES:
Overall Survival（OS） | Up to ~36 months
Overall response rate（ORR） | Up to ~24 months
Clinical benefit rate（CBR） | Up to ~24 months
Disease control rate（DCR） | Up to ~24 months
Duration of Response（DOR） | Up to ~24 months
Safety and Tolerability：the incidence and severity of treatment emergent adverse events (TEAEs) and serious adverse events (SAEs) | Up to ~24 months
PK metrics：plasma concentration of sirolimus | Up to ~24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trials Information Group, Shijiazhuang, Hebei, China